CLINICAL TRIAL: NCT01448200
Title: A Phase 1 Dose-Ranging Study to Assess the Safety, Pharmacokinetics and Antiviral Efficacy of PPI-668 in Healthy Volunteers and Patients With HCV Genotype-1 Infection
Brief Title: A Phase 1 Study of PPI-668 in Healthy Volunteers and Patients With Hepatitis C Virus (HCV) Genotype 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Presidio Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PPI-668-101
Record Dates: First submitted 2011-10-05; First posted 2011-10-07 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Hepatitis C, Chronic
Keywords: hepatitis C; NS5A inhibitor; Phase 1; genotype-1; genotype-2; genotype-3
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — ravidasvir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Part I: single dose escalation in healthy volunteers (Experimental): There will be three sequential single dose cohorts:
  Cohort A: PPI-668 dose D1 or placebo
  Cohort B: PPI-668 dose D2 or placebo
  Cohort C: PPI-668 dose D3 or placebo
  Interventions: Drug: PPI-668; Drug: Placebo
- Part I: multiple dose administration to healthy volunteers (Experimental): Upon completion of the single dose escalation phase, an additional cohort will receive repeat doses:
  Cohort D: highest well-tolerated dose from Cohorts A-C or placebo once daily for five days
  Interventions: Drug: PPI-668; Drug: Placebo
- Part II: multiple dose escalation in HCV subjects (Experimental): Upon completion of Part I, there will be 3, and potentially 4, sequential cohorts of HCV patients:
  Cohort E (genotype-1): PPI-668 dose E1 or placebo
  Cohort F (genotype-1): PPI-668 dose E2 or placebo
  Cohort G (genotype-1): PPI-668 dose E3 or placebo
  Cohort H (genotype-1): if necessary for dose-response assessment; dose to be determined
  Cohort I (genotype-2 or -3): PPI-668 dose E4 or placebo
  Interventions: Drug: PPI-668; Drug: Placebo

INTERVENTIONS:
Drug: PPI-668 — capsules
Drug: Placebo — capsules

SUMMARY:
PPI-668 is an antiviral agent (a hepatitis C NS5A inhibitor) that is being developed as a potential treatment for hepatitis C virus infection. This study is being done to assess the safety and tolerance of PPI-668 when given to healthy volunteers for up to 5 days (Part I of the study) and to hepatitis C patients for up to 3 days (Part II). In addition, the study will assess how much PPI-668 is absorbed into the bloodstream. In Part II, the effect of PPI-668 on the amount of hepatitis C virus in patients' bloodstream (serum HCV RNA levels) also will be assessed.

ELIGIBILITY:
In order to participate in the study, volunteers for Part I and patients for Part II must meet all of the following key entry criteria, as well as other entry criteria specified in the full protocol:

Key Inclusion Criteria

1. Male or female, between 18 and 65 years of age. Female patients must be surgically sterile or two years post-menopausal.
2. Body Mass Index (BMI) 18 - 35 kg/m2
3. In good health, in the judgment of the Principal Investigator
4. Able and willing to comply with all protocol requirements and to sign an informed consent.

Key Exclusion Criteria:

1. Seropositive for HIV antibody, or HBV surface antigen (HBsAg) at Screen. Volunteer subjects for Part I must also be negative for HCV antibody.
2. Any medical condition that may interfere with the absorption, distribution or elimination of study drug (PPI-668), or with the clinical and laboratory assessments in this study.
3. Poorly controlled or unstable hypertension; or sustained systolic BP > 150 or diastolic BP > 95 at Screen.
4. History of Diabetes Mellitus treated with insulin or hypoglycemic agents
5. History of alcohol abuse or illicit drug use which, in the investigator's judgment, could interfere with a patient's compliance, with the protocol requirements or with the safety or efficacy assessments of the study
6. History of malignancy unless the malignancy has been in complete remission and without additional medical or surgical interventions during the preceding three years
7. No clinically significant laboratory abnormalities at Screen for healthy volunteers in Part I. For Screen laboratory parameters for HCV patients in Part II, refer to the 'Additional Criteria for HCV Patients' below.

Additional Key Entry Criteria for HCV patients (Part II):

1. Clinical diagnosis of chronic hepatitis C, documented by:

   1. Clinical findings compatible with chronic hepatitis C, and absence of other known liver disease
   2. Seropositive for HCV antibody or HCV RNA at least once previously, and at Screen
   3. Serum HCV RNA > 5 log10 IU/mL at Screen, by the PCR assay at the central study laboratory
   4. HCV genotype-1 (1a or 1b, or non-subtypable genotype-1), or HCV genotype-2a or genotype-3a
2. ALT must be <5 x ULN at screen
3. No previous treatment with interferon, pegIFN, or ribavirin for genotype-1 patients
4. No history of signs or symptoms of decompensated liver disease
5. Any of the following laboratory values at Screening will be exclusionary for study participation:

   * Hgb <11 g/dL in women or 12 g/dL in men.
   * White blood cell count < 4,000/mm3.
   * Absolute neutrophil count (ANC) < 1800 per mm3.
   * Platelet count < 100,000 per mm3.
   * Serum creatinine >ULN at the central study laboratory.
   * Serum albumin < 3.4 g/dL.
   * Total bilirubin > 2.0 mg/dL
   * Clinically significant abnormality in the electrocardiograms (ECGs) at Screen

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2011-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability, as measured by clinical adverse events and laboratory assessments | Part I, up to day 12; and Part II, up to day 17

SECONDARY OUTCOMES:
PPI-668 plasma levels | Part I, up to day 12; and Part II, up to day 17
serum HCV RNA levels | Part II, up to day 17

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel Brown, M.D., Study Director — Presidio Pharmaceuticals, Inc.
Locations (7):
- United States (4):
  - Investigational site, Costa Mesa, California
  - Investigational site, Sacramento, California
  - Investigational site, San Francisco, California
  - Investigational Site, San Antonio, Texas
- Investigational site, Canberra, Australia
- New Zealand (2):
  - Investigational site, Auckland
  - Investigational site, Christchurch